CLINICAL TRIAL: NCT01407783
Title: Systems of Care for New Moms: Integrating Depression Treatment
Acronym: NUMOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nurses for Newborns Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R34MH083085-02 (NIH)
Record Dates: First submitted 2011-07-28; First posted 2011-08-02 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Post-partum Depression
Keywords: Post-partum depression; Low-income mothers; home nurse visitation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Solving Tools (Experimental): The home visitation nurse will teach and utilize the problem solving tools to help low-income depressed mothers. It is a brief treatment with the a non-pathologizing intervention being done in 4-8 sessions.
  Interventions: Behavioral: Problem Solving Tools (PST)
- Enhanced Referral (No Intervention)

INTERVENTIONS:
Behavioral: Problem Solving Tools (PST) — The problem solving tools was chosen as the depression treatment because it is well suited for use by non-mental health professionals and for in-home treatment. It is also a brief treatment (4-8 sessions) that takes a non-pathologizing approach.
  Other Names: Problem Solving Therapy
  Arms: Problem Solving Tools

SUMMARY:
NUMOMS involves collaboration between Nurses for Newborns Foundation and Washington University in St. Louis. This study explores the co-location of depression treatment within nurse home visitation and the organizational changes needed to maintain access to evidence-based treatment. Problem Solving Tools (PST) was chosen as the depression treatment because it is well suited for use by non-mental health specialists and for in-home treatment. It is also a brief treatment (4-8 sessions) takes a non-pathologizing approach.

DETAILED DESCRIPTION:
NUMOMS involves collaboration between Nurses for Newborns Foundation and Washington University in St. Louis. This study explores the co-location of depression treatment within nurse home visitation and the organizational changes needed to maintain access to evidence-based treatment. Problem Solving Tools (PST) was chosen as the depression treatment because it is well suited for use by non-mental health specialists and for in-home treatment. It is also a brief treatment (4-8 sessions) takes a non-pathologizing approach.

In the first part of the study we will gather information from women and their providers to determine what system and treatment modifications are needed to effectively deliver acceptable depression treatment in home visitation programs. Based on this information, a panel of local and national experts will provide advice on decisions regarding the intervention adaptation. Once these adaptation decisions are made a small group of experts will adapt a PST manual for use in home visitation.

In the second phase of the NUMOMS study we will carry out a small two-arm randomized trial comparing the effectiveness, acceptability, and practicality of PST provided by home visitation RNs versus usual care (referral to mental health specialty care).

Significantly, NUMOMS has the potential to provide home visitation agencies with a viable means of access to effective and acceptable depression treatment for mothers in the face of policy mandates for depression screening.The specific aims are to:

1. Adapt PST for implementation in nurse home visitation programs.

   1. Examine internal (organization and client level) and external (community and policy level) factors that may impact upon PST adaptation and delivery in nurse home visitation.
   2. Build protocols for targeting depression treatment to the woman's symptom severity and patient preferences.
   3. Develop and routinize protocols for supervision, clinical consultation, and risk assessment for PST provided by nurse home visitors.
   4. Modify protocols and systems for client tracking and outcomes.
2. Implement a two-arm randomized pilot study comparing: PST provided by non-mental health home visitation nurses and referral for treatment (Care as Usual).

   1. Compare outcomes on the Beck Depression Inventory, the Patient Health Questionnaire-9, and Parenting Stress Index for women treated with PST by non-specialty RNs and Care as Usual.
   2. Track pathways and barriers to care for women referred to mental health specialty care or primary care for medications.
   3. Develop an R01 for a full scale randomized controlled trial using data on effect sizes and addressing organizational issues, infrastructure needs, and treatment refinements.

ELIGIBILITY:
Inclusion Criteria:

* Depressed as indicated by Edinburgh Postpartum Depression Scale or Clinical Checklist
* NFNF client from a certain zip code
* Either pregnant or have a child under the age of 12 months in the home

Exclusion Criteria:

* Under the age of 18
* Severe Mental Illness
* Chemical Dependency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | baseline, 6months and 12 months post treatment
  Measure the reduction of post partum depression after intervention at 6 months and 12 months post treatment.
BDI-II | baseline, 6months &12 months post treatment
  Measure the reduction of post partum depression after intervention at 6 months and 12 months post treatment.

SECONDARY OUTCOMES:
Qualitative Interview | 1 month post treatment
  Questions asking the participants their feelings about the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Zayas, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University and Nurses for Newborns Foundations, St Louis, Missouri, United States